CLINICAL TRIAL: NCT02746458
Title: REPAIR: Rehabilitation Enhanced by Partial Arterial Inflow Restrictions
Brief Title: Rehabilitation Enhanced by Partial Arterial Inflow Restrictions
Acronym: REPAIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-15-2-0067
Record Dates: First submitted 2016-04-07; First posted 2016-04-21 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Closed Femur Fracture
Keywords: Blood Flow Restriction; Muscle Weakness; Physical therapy techniques; closed femoral fracture injuries
MeSH Terms: conditions — Muscle Weakness | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Physical Therapy (No Intervention): This group will receive the standard of care physical therapy program for 6 weeks.
- Blood Flow Restriction Plus Standard of Care Physical Therapy (Experimental): This group will receive the same standard of care physical therapy program for 6 weeks plus blood flow restriction.
  Interventions: Other: Blood Flow Restriction; Device: Delfi PTSII Tourniquet System

INTERVENTIONS:
Other: Blood Flow Restriction — Brief and intermittent blood flow restriction via a Delfi PTSII Tourniquet System will be used during physical therapy.
  Arms: Blood Flow Restriction Plus Standard of Care Physical Therapy
Device: Delfi PTSII Tourniquet System
  Arms: Blood Flow Restriction Plus Standard of Care Physical Therapy

SUMMARY:
The Rehabilitation Enhanced by Partial Arterial Inflow Restriction (REPAIR) Study will be conducted in a patient population of individuals recovering from a traumatic diaphyseal fracture of the femur. Although the intervention can be used for any patient with muscle weakness following trauma, the persistent thigh weakness that follows a femur fracture provides a perfect model for evaluating the effectiveness of the REPAIR protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-55 inclusive
2. Admitted to one of the participating clinical centers for operative treatment of a closed diaphyseal femur fracture with one of the following OTA codes: 32A, 32B or 32C (treated with an IM Nail).

Exclusion Criteria:

1. Open diaphyseal femur fracture (except low velocity gunshot wounds) or severe crushing injuries to study limb.
2. Additional fracture, dislocations or soft tissue injuries to the study limb that would compromise the ability to weight bear as tolerated and initiate PT within 28 days of definitive fixation.
3. Any fractures, dislocations or soft tissue injuries to the contralateral limb or pelvis that would compromise the ability to weight bear as tolerated and initiate PT within 28 days of definitive fixation.
4. Any treatment of the study injury in either group that would preclude application of the tourniquet cuff (e.g. vascular reconstruction, wound, flap, or skin graft).
5. Injuries to other body systems (or other medical conditions) that would preclude the ability to weight bear as tolerated and initiate PT within 28 days of definitive fixation (e.g. spinal cord deficit; severe traumatic brain injury).
6. Use of blood flow restriction (BFR) at any time between treatment and the start of physical therapy for the study.
7. Non-ambulatory pre-injury.
8. Morbidly obese (BMI > 40).
9. History of Peripheral Artery Disease and/or Peripheral Vascular Disease (PAD/PVD).
10. Current or history of venous thromboembolism.
11. Impaired circulation or peripheral vascular compromise.
12. Previous revascularization at the study injury site.
13. Extremities with dialysis access.
14. Current diagnosis of acidosis.
15. Diagnosis of sickle cell anemia.
16. Current infection of the study injury.
17. Current tumor (malignant or benign) distal to study injury and future tourniquet placement.
18. Current use of medications or supplements that are known to increase clotting risk.
19. Diagnosis of severe hypertension (blood pressure of 180/110).
20. Skin grafts in which all bleeding points must be readily distinguished.
21. Secondary or delayed surgical procedures to study injury after immobilization.
22. Vascular grafting to the study injury.
23. History of lymphotomies.
24. Current diagnosis of cancer.
25. Unable to speak either English or Spanish.
26. Severe problems with maintaining follow-up (e.g. patients who are prisoners, homeless at the time of injury, who are intellectually challenged without adequate family support, or have document psychiatric disorders).
27. Unable to provide informed consent.
28. Patient has not been cleared to start physical therapy at the time of consent.
29. Patient is pregnant.
30. Patient received BFR between date of injury and start of Physical Therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Knee Strength measured using a stabilized hand held dynamometer | up to 6 months
  Knee strength will be measured using a stabilized hand held dynamometer in both the injured and uninjured legs.
Muscle Volume assessed using mid-thigh girth circumference measurement | up to 6 months
  Muscle volume will be assessed using mid-thigh girth circumference measurements.

SECONDARY OUTCOMES:
Strength | up to 6 months
  Strength will be measured using the sit to stand test.
Speed | up to 6 months
  Speed will be evaluated using the self selected walking speed.
Speed | up to 6 months
  Speed will be evaluated using the 40 yard shuttle run.
Posture Stability | Change in Functional Performance Measures at 3 months and 6 months
  Postural stability will be evaluated using the single leg stance.
Agility | up to 6 months
  Agility will be measured using the 4 step square test.
Agility | up to 6 months
  Agility will be measured using the Illinois Agility Test.
Physical Function | up to 1 year
  Physical Function will be evaluated by the Patient Reported Outcomes Measurement Information System physical function questionnaire.
Depression evaluated with a depression questionnaire | up to 1 year
  Depression will be evaluated by the Patient Reported Outcomes Measurement Information System depression questionnaire.
Anxiety evaluated with an anxiety questionnaire | up to 1 year
  Anxiety will be evaluated by the Patient Reported Outcomes Measurement Information System anxiety questionnaire.
Sleep Disturbance evaluated with a sleep disturbance questionnaire | up to 1 year
  Sleep Disturbance will be evaluated by the Patient Reported Outcomes Measurement Information System sleep disturbance questionnaire.
Psychological outcome-Post Traumatic Stress (PTSD) measured using the standard PTSD Checklist (PCL) | up to 1 year
  PTSD will be measured using the standard PTSD Checklist (PCL).
Return to Work and Work Productivity measured using the Work Productivity and Activity Impairment (WPAI) questionnaire | up to 1 year
  Work productivity will be measured using the Work Productivity and Activity Impairment (WPAI) questionnaire.
Pain evaluated with a Pain Inference scale | up to 1 year
  Pain will be evaluated by the Patient Reported Outcomes Measurement Information System Pain Inference scale.
Satisfaction with Care and Recovery assessed using the MedRisk Instrument for Measuring Patient Satisfaction with Physical Therapy Care (MRPS) | 3 months
  This will be assessed using the MedRisk Instrument for Measuring Patient Satisfaction with Physical Therapy Care (MRPS).
Fracture Healing | up to 1 year
  Fracture healing will be determined by clinical examinations.
Fracture Healing | up to 1 year
  Fracture healing will be determined by radiographic examinations.
Complications | up to 1 year
  The presence of all limb related complications will be recorded prospectively at each follow up visit, and categorized according to type, date diagnosed, severity, treatment and relation to the study injury.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reider, PhD, Study Director — Major Extremity Trauma Research Consortium Coordinating Center; Daniel J Stinner, MD, Principal Investigator — San Antonio Military Medical Center; Ellen J MacKenzie, PhD, Principal Investigator — Major Extremity Trauma Research Consortium Coordinating Center
Locations (8):
- United States (8):
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Barnes Jewish Hospital, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - MetroHealth, Cleveland, Ohio
  - University of Texas Health Science Center at Houston, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No